CLINICAL TRIAL: NCT03148288
Title: Vitamin D Supplementation in IBS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 2017P000133
Record Dates: First submitted 2017-05-09; First posted 2017-05-10 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Irritable Bowel Syndrome; Vitamin D Deficiency; Abdominal Pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Vitamin D Deficiency; Abdominal Pain | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D supplementation (Experimental): 4000IU Vitamin D qd
  Interventions: Dietary Supplement: Vitamin D
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — VItamin D
  Arms: Vitamin D supplementation
Dietary Supplement: placebo — placebo
  Arms: placebo

SUMMARY:
Irritable bowel syndrome (IBS) is a very common functional gastrointestinal disorder affecting nearly 20% of the North American population. IBS is characterized by chronic abdominal, associated with a change in bowel frequency and or consistency that lack a known structural or anatomic explanation. Current treatment for IBS is primarily symptom-based. However over a third of patients with IBS fail to respond to currently available therapies.

The prevalence of vitamin D deficiency/insufficiency is estimated in over a billion people world-wide . Vitamin D has potential mechanisms not only in the balance of calcium and bone homeostasis, but also a key modulator of the immune system. Vitamin D receptors (VDRs) are located on all nucleated cells including the GI tract. Thus far, there is already accumulating evidence for a role for vitamin D supplementation in inflammatory bowel disease (IBD). A recent systematic review suggested there may be benefits of vitamin D supplementation in IBD.

Vitamin D insufficiency is widespread in patients with IBS and there is a positive association between vitamin D status and quality of life. To date, there is no US trial examining the effect of vitamin d supplementation on IBS symptoms and quality of life in patients with IBS.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent and understand the nature of the study sufficiently to allow completion of all study assessments.
2. Be ambulatory, community dwelling, 18 to 80 years, inclusive
3. Meet Rome IV diagnostic criteria for IBS
4. Have IBS of at least "moderate" severity, i.e., have a score on the IBS-SSS of > 175 (0-500) at the baseline visit (Visit 1)
5. If the patient is on medications which affect the gastrointestinal tract or visceral sensation (e.g., tricyclic antidepressants, fiber, antispasmodics, etc.) they must be on a stable dose for at least 1 month prior to entering the study and for the duration of the study.

Exclusion Criteria:

1. Have a history of intractable IBS, defined as continuous, unremitting and severe abdominal pain.
2. Be pregnant or lactating.
3. Have an established diagnosis of any concomitant bowel disturbance that would interfere with the assessment of efficacy or safety in the study (e.g., Hirschsprung's disease, inflammatory bowel disease, celiac disease).
4. Report warning symptoms (i.e., rectal bleeding, weight loss >10%, iron deficiency anemia, etc.) otherwise not explained
5. Have undergone previous abdominal surgery (with the exception of uncomplicated appendectomy, cholecystectomy, hysterectomy, or polypectomy > 6 months prior to enrollment).
6. Have a history of metabolic or inflammatory disease that may affect bowel motility (e.g., inflammatory bowel disease, celiac, sarcoidosis, connective tissue disease, amyloidosis, or poorly controlled hypo/hyperthyroidism).
7. Have a history of significant concomitant psychiatric, neurological, metabolic, hepatic, renal, infectious, hematological, cardiovascular, gastrointestinal, or pulmonary illness. If there is a history of such disease but the condition has been stable for more than one year and is judged by the Investigator not to interfere with the patient's participation in the study, the patient may be included. Staff will document such cases.
8. Have a history of drug, excluding nicotine or caffeine, or alcohol abuse within 2 years of entry into the study
9. Exhibit abnormalities on physical examination, have abnormal vital signs, or clinical laboratory values, unless these abnormalities are judged to be clinically insignificant by the Investigator. Such cases will be noted.
10. Active laxative abuse.
11. Unable or unwilling to cooperate with the study protocol or considered by the Investigator to be unsuitable for the study.
12. Currently taking Vitamin D supplements
13. Diagnosis of osteoporosis
14. Currently bisphosphonate medications
15. Those who taking medication known to interfere with Vit D

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome - Symptom Severity Scale (IBS-SSS) | 12 weeks
  VAS on abdominal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No